CLINICAL TRIAL: NCT02763709
Title: Evaluation of Pediatric Critical Illness Neuropathy/Myopathy in Pediatric Intensive Care Unit
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Ananthanarayanan, Senior resident, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: PEDCIMP2016
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Critical Illness Polyneuropathy
MeSH Terms: conditions — Polyneuropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cases: Children admitted in Pediatric ICU for more than 24 hours with Pediatric Risk of Mortality (PRISM) score III > 20

SUMMARY:
Intensive Care Unit Acquired Weakness(ICUAW) encompasses a spectrum of disorders characterized by generalized weakness developing after the onset of critical illness. Pediatric data on the incidence of ICUAW is restricted to isolated case reports and case series of no more than five children. Critical illness polyneuropathy is characterized by reduction in compound motor action potential or sensory nerve action potential or both with preserved conduction velocity on electrophysiological studies. These findings can occur very early prior to the onset of clinical features. Given the dearth of data in children on the subject, this study has been planned to evaluate the incidence of critical illness associated polyneuropathy /myopathy in severely sick children admitted.

DETAILED DESCRIPTION:
Materials and Methods

Study Setting: Pediatric Intensive Care Unit, Advanced Pediatric Centre, Postgraduate Institute of Medical Educational Research

Study Period: Jan 2016 to Dec 2016

Study design: Prospective Cohort Study

Study Population: Children of 2 years to 12 years of age

Study flow

All consecutive patients between the age group 2 years to 12 years admitted in Pediatric Intensive Care Unit (ICU) in Advanced pediatric Centre with PRISM score of more than 20 will screened for inclusion in the study.Those found eligible would be included after an informed consent. Baseline clinical and demographic profile will be recorded on a proforma.

Entry Examination

Clinical Evaluation

It would include history and examination. A clinical evaluation will be performed at the time of patient recruitment and then daily till discharge from ICU. It would also include assessment of the Glasgow Coma Scale, the Sequential Organ System Failure score (SOFA) and tendon reflexes. The muscle strength of the main muscle groups will be graded using the Medical Research Council (MRC) scale in cooperative children.

* Upper Extremity: Wrist Extension, Elbow Flexion, Shoulder Abduction
* Lower Extremity: Ankle Dorsiflexion, Knee Extension, Hip Flexion

Scoring & Interpretation:

* Maximum Score: 60 (4 Limbs, Maximum of 15 Points Per Limb) = Normal
* Minimum Score: 0 = Quadriplegia

Severity of multi organ failure will be assessed by mean SOFA scores during ICU stay, highest SOFA scores and sum of 28-day total SOFA scores in every patient.

The total dose and duration of drug therapy like steroids, muscle relaxants, sedatives and inotropes will also be entered. Laboratory parameters like serum creatine kinase, albumin, total protein, serum electrolytes and plasma blood glucose will also quantified.

Electrophysiological Evaluation

Twenty fours after admission, entry examination in the form of complete nerve conduction study from 4 motor nerves (median, ulnar, tibial and common peroneal nerve) and 2 sensory nerves (median and sural nerve) will be performed. These will consist of Compound Motor Action Potential(CMAP) measurement from motor nerves and Sensory Nerve Action Potential (SNAP) assessment from sensory nerves. Before the electrophysiological tests, heat packs will be applied to the skin if its temperature is below 33°C.

Serial Examination

Following the detailed entry evaluation, daily simplified electrophysiological tests in the form of conduction velocity and amplitude of the sural SNAP and common peroneal CMAP in one leg using surface electrode stimulation and recording electrodes will be assessed. To minimize artifacts, the same electrode site will be marked and similar size electrode will be used for each patient on a daily basis. A 25% decrease from baseline SNAP and CMAP measured at ICU admission will be taken as the minimum consistently detectable reduction.If SNAP or CMAP decreases by more than 25% on two consecutive days, a complete electrophysiological test will be performed. Complete electrophysiological testing includes nerve conduction study and electromyography.Electromyography will be recorded using a coaxial needle electrode in the tibialis anterior and first dorsal interossei.If the complete electrophysiological test is consistent with critical illness weakness, complete weekly tests will replace daily tests until ICU discharge.

ELIGIBILITY:
Inclusion Criteria:

* Children admitted in Pediatric Intensive Care Unit for more than 24 hours
* Pediatric Risk of Mortality (PRISM) score III > 20

Exclusion Criteria:

* Previous (Eg: Diabetes Mellitus, Systemic Lupus Erythematosus, Dermatomyositis, Spinal Muscular Atrophy) or current neuromuscular disorder (e.g Guillian Barre Syndrome, snake bite, myositis)
* Use of drugs causing neuromuscular blockade
* Bilateral Lower limb disorders precluding Nerve Conduction Study or ElectroMyoGraphy (Gross edema, fractures, amputation, plaster casts, open wounds, infections)
* Children with abnormal electrophysiological studies at baseline examination will be excluded

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children admitted in Pediatric Intensive Care Unit for more than 24 hours with a Pediatric Risk of Mortality (PRISM) score III > 20
Sampling Method: Probability Sample
Enrollment: 97 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Pediatric critical illness polyneuropathy/myopathy | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Naveen Sankhyan, DM, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh; Pratibha Singhi, MD, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- PGIMER, Chandigarh, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kasinathan A, Sharawat IK, Singhi P, Jayashree M, Sahu JK, Sankhyan N. Intensive Care Unit-Acquired Weakness in Children: A Prospective Observational Study Using Simplified Serial Electrophysiological Testing (PEDCIMP Study). Neurocrit Care. 2021 Jun;34(3):927-934. doi: 10.1007/s12028-020-01123-x. Epub 2020 Oct 7. PMID 33025545